CLINICAL TRIAL: NCT03681106
Title: Efficacy of Kinesio® Tex Taping on Edema and Early Functional Outcome of Post Total Knee Replacement Patients: a Randomized-controlled Trial
Brief Title: Kinesio® Tex Taping for Post Total Knee Replacement Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the health crisis triggered by the COVID-19 pandemic and the consequent sanitary-organizational arrangements set up for its contrast it was necessary to interrupt the study before reaching the established sample size.
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kinesiotaping
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Total Knee Arthroplasty; Kinesiotaping; Neuro taping; Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Masking Description: Randomization list has been already generated but will not be available to the recruiters to avoid allocation bias.
  Statistician that will handle the data analysis will not know which group is the interventional and which group is the control.
  We were not able to mask the using of tape to the patients or the investigators because it is an evident treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape (Experimental): Kinesio Tex taping treatment for 10 days + usual care
  Interventions: Device: Kinesio Tex
- Control (No Intervention): usual care

INTERVENTIONS:
Device: Kinesio Tex — Kinesio Tex tape on the operated limb
  Arms: Kinesiotape

SUMMARY:
This study is designed to better understand the effect of Kinesio Taping applied using the Neurotaping technique on patients who underwent total knee arthroplasty surgery. Patients will be randomized in two groups: in the first group patients will follow a protocol of usual rehabilitation, while the second group will do the same but add the Kinesio Taping application. Main outcome will be the effect on edema, secondary outcome the effect on functionality after 13 days post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Program of total knee replacement;
* Signing and accepting informed consent.

Exclusion Criteria:

* pre-operative Barthel Index score < 70;
* program of revision of total knee replacement;
* grade III-IV heart failure;
* grade III-IV kidney failure;
* hypersensitive skin or intolerance to taping;
* Active cutaneous infection or open skin lesion on the sites of taping positioning;
* Body Mass Index > 34,9;
* Pregnant women;
* Not accepting informed consent;
* Impossibility to follow usual rehabilitation treatment.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Knee circumference | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  Difference between pre-operative knee circumference and 13th post-operative day knee circumference expressed in cm

SECONDARY OUTCOMES:
Timed Up and Go test | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  Functional test
10 meters walking test | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  Functional test
Barthel Index | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  Autonomy outcome
Functional Independence Measure | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  Autonomy outcome
Knee range of motion | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  Flexion/extension passive/active range of motion of operated knee
Thigh circumference | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  Thigh circumference expressed in cm
Leg circumference | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  Leg circumference expressed in cm
Ankle circumference | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  Ankle circumference expressed in cm
Pain Visual Analogue Scale | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  The Pain Visual Analogue Scale scale consists of a straight line, 10 cm long, printed on a white sheet, the endpoints, 0 and 10, defining respectively "no pain at all" and "pain as bad as it could be". The patient must mark the line to indicate his perception of his level of pain at that time.
R0 measured using bioimpedance | pre-operative, 3rd post-operative day, 7th post operative day, 13th post-operative day
  body impedance

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Negrini, MD, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williams S, Whatman C, Hume PA, Sheerin K. Kinesio taping in treatment and prevention of sports injuries: a meta-analysis of the evidence for its effectiveness. Sports Med. 2012 Feb 1;42(2):153-64. doi: 10.2165/11594960-000000000-00000. PMID 22124445
- [Background] Morris D, Jones D, Ryan H, Ryan CG. The clinical effects of Kinesio(R) Tex taping: A systematic review. Physiother Theory Pract. 2013 May;29(4):259-70. doi: 10.3109/09593985.2012.731675. Epub 2012 Oct 22. PMID 23088702
- [Background] Bade MJ, Stevens-Lapsley JE. Restoration of physical function in patients following total knee arthroplasty: an update on rehabilitation practices. Curr Opin Rheumatol. 2012 Mar;24(2):208-14. doi: 10.1097/BOR.0b013e32834ff26d. PMID 22249349
- [Background] Wozniak-Czekierda W, Wozniak K, Hadamus A, Bialoszewski D. Use of Kinesiology Taping in Rehabilitation after Knee Arthroplasty: a Randomised Clinical Study. Ortop Traumatol Rehabil. 2017 Oct 31;19(5):461-468. doi: 10.5604/01.3001.0010.5828. PMID 29154230
- [Background] Donec V, Krisciunas A. The effectiveness of Kinesio Taping(R) after total knee replacement in early postoperative rehabilitation period. A randomized controlled trial. Eur J Phys Rehabil Med. 2014 Aug;50(4):363-71. Epub 2014 May 13. PMID 24819349